CLINICAL TRIAL: NCT07199049
Title: Monitoring Eyelid Reflex, Eye Movements, and Pupil Responses in Patients Undergoing General Anesthesia: Neuro-Mimic Indicators of Anesthesia Depth
Brief Title: Neuro-Mimic Indicators of Anesthesia Depth During General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: NEURO3419
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: General Anesthesia; Intraoperative Awareness; Eye Movements
Keywords: Anesthesia, General; Awareness, Intraoperative; Pupillary Reflex; Eye Movements; Reflex, Blink (Eyelid Reflex)
MeSH Terms: conditions — Intraoperative Awareness | interventions — Eye Movements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neuro-Mimic Observation Protocol — Observation of eyelid reflex, eye movements, and pupil responses at three standardized intraoperative time points (after induction, during skin incision, and mid-surgery). Parameters will be recorded alongside BIS values without any intervention, device application, or additional risk to patients.
  Other Names: Eyelid Reflex Monitoring; Eye Movement Observation; Pupil Diameter Assessment

SUMMARY:
This prospective observational study will evaluate neuro-mimic indicators of anesthesia depth, including eyelid reflex, eyeball movements, and pupil responses, in patients undergoing elective surgery under general anesthesia. Sixty adult patients will be observed at three standardized time points: after induction, during skin incision, and mid-surgery. All parameters will be recorded alongside bispectral index (BIS) monitoring. The study aims to determine whether these observable signs correlate with anesthesia depth, contribute to early detection of intraoperative awareness, and provide a basis for developing non-invasive depth monitoring systems.

DETAILED DESCRIPTION:
Accurate assessment of anesthesia depth is essential to ensure patient safety and reduce the risk of intraoperative awareness. Current technological monitoring tools such as BIS do not always provide sufficient reliability. Neuro-mimic indicators, including eyelid reflex, spontaneous and stimulus-related eye movements, and pupil responses, may offer additional insights into anesthesia depth. This observational, prospective, non-interventional study will enroll 60 adult patients (aged 18-65, ASA I-III) scheduled for elective abdominal surgeries lasting 1-3 hours under general anesthesia at Başakşehir Çam and Sakura City Hospital. Observations will be performed at three intraoperative stages: post-induction, skin incision, and mid-surgery. Parameters include palpebral reflex, eyeball position and movement, and pupil diameter, all systematically documented alongside BIS values. The primary endpoint is the change in pupil diameter across three time points. Secondary outcomes include the presence or absence of eyelid reflex, eye movements, and their correlations with BIS values. Data will be analyzed using repeated measures ANOVA, McNemar test, correlation analyses, and appropriate non-parametric tests where necessary. The study is entirely observational and involves no additional interventions or risks for patients. Results may provide evidence for the integration of observable physiological signs into anesthesia monitoring practice and contribute to the development of contactless depth monitoring systems.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients aged 18-65 who will undergo elective abdominal surgery (e.g., cholecystectomy/gastrectomy/colorectal surgery/prostatectomy/hysterectomy, etc.) under general anesthesia, with a planned duration of 1-3 hours.
* Patients whose eye area is left uncovered and who are in a position suitable for observation
* Patients who have signed the informed consent form
* Patients with an ASA score of I-III

Exclusion Criteria:

* Patients undergoing surgical procedures in the head, neck, or face region (e.g., ENT, eye, jaw surgery, neurosurgery, thyroid/parathyroid)
* Patients whose eye area must be completely covered with a sterile drape
* Patients with an ASA score of IV or higher
* Individuals with neurological disorders and impaired pupil response, patients who have previously undergone eye trauma or surgery and cannot undergo pupil evaluation
* Patients who are unable to communicate and cannot provide informed consent
* Emergency surgeries (e.g., appendectomy/ileus/gastrointestinal perforation/cesarean section/gunshot wounds/stab wounds/multiple trauma/traffic accidents, etc.)
* Individuals who have previously been included in this study (to prevent repeated inclusion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years, ASA physical status I-III, undergoing elective abdominal surgery under general anesthesia at Başakşehir Çam and Sakura City Hospital will be included. Eligible patients must have the eye area uncovered and in a position suitable for observation, with surgery expected to last 1-3 hours. Both male and female patients will be enrolled. Head, neck, and eye surgeries or cases requiring full draping of the eye area will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in pupil diameter during general anesthesia | Intraoperative period (observations at induction, incision, and mid-surgery).
  Pupil diameter (mm) will be measured and compared at three intraoperative stages: after induction and intubation, during skin incision, and mid-surgery. The change over time will be analyzed as an indicator of anesthesia depth.

SECONDARY OUTCOMES:
Presence or absence of eyelid reflex at different anesthesia stages | Intraoperative period (induction, incision, mid-surgery).
  Eyelid reflex (palpebral reflex) will be assessed as present or absent at three intraoperative stages and analyzed in relation to anesthesia depth.
Eye position and movements during anesthesia | Intraoperative period (induction, incision, mid-surgery).
  Eyeball position (central, upward, downward, eccentric) and spontaneous movements will be observed and documented at three time points. Changes will be evaluated as neuro-mimic indicators of anesthesia depth.
Correlation of neuro-mimic indicators with BIS values | Intraoperative period (induction, incision, mid-surgery).
  Observed eyelid reflex, eye movements, and pupil responses will be correlated with simultaneously recorded BIS values to explore associations with anesthesia depth.
Early indicators of intraoperative awareness | Intraoperative period.
  The relationship between observed neuro-mimic responses (eyelid reflex, eye movements, pupil diameter) and intraoperative awareness risk will be evaluated descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ozcan, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns. Only summary-level data and aggregated results will be published in scientific journals or presented at conferences.

REFERENCES:
- [Background] Ben Barak-Dror O, Hadad B, Barhum H, Haggiag D, Tepper M, Gannot I, Nir Y. Touchless short-wave infrared imaging for dynamic rapid pupillometry and gaze estimation in closed eyes. Commun Med (Lond). 2024 Aug 6;4(1):157. doi: 10.1038/s43856-024-00572-1. PMID 39107497
- [Background] Singh A, Akhileshwar, Kumar N, De RR, Bahadur R, Shekhar S. The Role of Pupillometry in the Assessment of Pain in Children Under General Anesthesia: A Prospective Single-Blinded Observational Study. Cureus. 2023 Aug 22;15(8):e43894. doi: 10.7759/cureus.43894. eCollection 2023 Aug. PMID 37753025
- [Background] Chaurasia S, Soni SL, Ganesh V, Ram J, Sukhija J, Chaurasia S, Takkar A. Tonic down-rolling and eccentric down-positioning of eyes under sevoflurane anesthesia without non-depolarizing muscle relaxant and its relationship with depth of anesthesia. Front Med (Lausanne). 2023 Jun 15;10:1029952. doi: 10.3389/fmed.2023.1029952. eCollection 2023. PMID 37396902
- [Background] Xing L, Xie H, Zhou X, Zhu J, Liu H. Ultrasound Measurement of Pupillary Dilation Reflex During Induction of General Anesthesia Using Sufentanil: A Randomized Controlled Trial. Med Sci Monit. 2025 Jun 23;31:e948209. doi: 10.12659/MSM.948209. PMID 40549665